CLINICAL TRIAL: NCT02988856
Title: Non-surgical Correction of Eye Lid Paralysis With External Magnet Systems
Brief Title: Magnetic Correction of Eye Lid Paralysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Houston (Other)
Responsible Party: Sponsor-Investigator, Kevin Houston, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-027H
Record Dates: First submitted 2015-10-01; First posted 2016-12-09 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Blepharoptosis; Lagophthalmos; Facial Paralysis
MeSH Terms: conditions — Blepharoptosis; Lagophthalmos; Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic lid system (Experimental): All participants will trial a commercially available device and an experimental magnetic device.
  Interventions: Device: Magnetic lid system

INTERVENTIONS:
Device: Magnetic lid system — Small externally mounted magnetic lid arrays are attached to the eye lid (s). Glasses with a second magnet system may be combined with the arrays depending on the lid condition. The device intends to facilitate eye opening and closing.
  Other Names: Magnetic Levator and Magnetic Orbicularis

SUMMARY:
Objective 1: Determine the safety and feasibility of externally mounted magnets for extended management of chronic eyelid movement disorders by measuring visual acuity and corneal and skin integrity and comfort over 8 weeks of wear. Objective 2: Collect preliminary data on the relative efficacy of external magnetic devices by comparing them to externally mounted lid weights and ptosis crutches using rating scales and video analysis of blink biomechanics.

DETAILED DESCRIPTION:
Two major types of eye lid movement disorders include lagophthalmos (incomplete closure of the eyelids) and blepharoptosis (incomplete opening of the eyelids). Both of these conditions occur because of a disruption in the normal agonist-antagonist neuro-muscular complex balance. Generally paralysis of the eyelid or facial muscles is responsible for the abnormality (the eyelids can close but not open, or open but not close). An external device, if able to generate an appropriately balanced force, could restore eyelid movement by performing the paralyzed function; for example, a ptotic (droopy) eyelid could be opened, and the functioning eyelid closure muscle could overcome the device's force. In prior work the investigators established proof-of-concept data demonstrating safety and efficacy for temporary management of ptosis up to 2 hour per day for 2 weeks. Preliminary data suggest similar safety for lagophthalmos. This study will expand on this preliminary work to examine longer wear times, home use, and feasibility for a wider range of eye lid disorders.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an eyelid movement disorder for at least one eye, moderate cognitive function or better defined as greater than or equal to 18 out of 30 on a pre-screening of the Mini-Mental State Exam, age 5 or older.

Exclusion Criteria:

* Absence of an eyelid movement disorder or presence of a corneal ulcer. Those with a corneal ulcer are at risk for permanent loss of vision and should be managed with proven methods. Age less than 5, Severe Cognitive impairment defined as Mini-mental score <18, behaviors consistent with delirium (combinations of disorientation, hallucinations, delusions, and incoherent speech), or lethargy. These individuals must be excluded since participation requires competent self-care, reliable responses and cooperation during fitting of the devices.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Houston, OD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Ophthalmology of Clinical Research Office, Mass Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Singh NK, Paschalis EI, Tomasi M, Rizzo JF, Houston KE. The boston blink-netic project: preliminary outpatient feasibility results (abstract). Optom Vis Sci 2016;93: E-abstract 16118.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnetic Lid System
Started | 11
Completed | 8
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Lid System
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Rating Scale of Skin Integrity
Description: Ratings at the beginning and end of treatment will be analyzed by calculating the mean and standard deviation of the skin erythema rating across all available time points. The outcome measure is the FDA scale, Assessing the Irritation and Sensitization Potential of Transdermal and Topical Delivery Systems for ANDAs Guidance for Industry. Range is 0 to 7 with higher numbers being worse skin erythema.
Time Frame: Baseline and up to 32 weeks
Population: Erythema rating in participants who had worn the MLP for 1 to 32 weeks. All the ratings each subject had across all their visits were averaged, and then a group average and std dev calculated.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnetic Lid System
Number analyzed (Participants) | 9
units on a scale | 0.3 (0.5)

2. Secondary Outcome: Count of Participants With Adverse Corneal Events Based on National Eye Institute Rating Scale
Description: Using the National Eye Institute Rating Scale (0 to 3 points with higher being more staining), cases where staining increased more than 2 points or if there was any ulceration, an adverse event was tabulated and summed for each participant over 1 up to 32 weeks of use, depending on how long the participant was followed.
Time Frame: Baseline and up to 32 weeks
Population: Participants with ptosis wearing the MLP for 1 or more weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Magnetic Lid System
Number analyzed (Participants) | 9
Participants | 1

3. Secondary Outcome: Change in Visual Acuity
Description: Visual acuity at 20ft before treatment and after 1 week or more. Difference between weekly acuity measures to baseline was calculated and averaged for each subject, and then a group mean and standard deviation calculated.
Time Frame: Baseline and up to 32 weeks
Population: Participants who wore the MLP for 1 week or more
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Magnetic Lid System
Number analyzed (Participants) | 7
LogMAR | 0.03 (0.08)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Magnetic Lid System
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Lid System (N=11)
Skin Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Corneal staining (Eye disorders) | 1 (1) — Increase in corneal staining over safety cutoff (>grade 2 increase)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT02988856/Prot_SAP_000.pdf